CLINICAL TRIAL: NCT05744570
Title: The Influence of the Anesthesiologists' Gender on Time Delay for Labor Epidural Anesthesia
Brief Title: Gender of Anesthesiologist and Time to Labor Epidural
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: TALW
Record Dates: First submitted 2023-02-10; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Labor Pain
Keywords: labor pain; epidural anesthesia; time delay
MeSH Terms: conditions — Labor Pain | interventions — Anesthesia, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male anesthesiologist: The anesthesiologist gender defined by first name
  Interventions: Procedure: Epidural anesthesia
- Female anesthesiologist: The anesthesiologist gender defined by first name
  Interventions: Procedure: Epidural anesthesia

INTERVENTIONS:
Procedure: Epidural anesthesia — Regional anesthesia for labor pain

SUMMARY:
The goal of this retrospective cohort study is to learn about wether the gender of the anesthetist affects time to epidural anesthesia (EDA) for laboring women . The main questions it aims to answer are:

1. Is there a gender difference in time to applying EDA
2. What is the mean waiting for EDA in laboring women in Sweden

Participants (anesthesiologists) will be reviewed according to the time from when the midwife asks for EDA to anesthesiologist register that it was in place

DETAILED DESCRIPTION:
In certain hospital in Sweden, a module on the most contemporary Obstetric chart system in Sweden allows for registration of time from request of EDA to applied EDA.Time of request is made by the midwife and the Tim of application is registered by the anesthesiologist. Not all hospitals makes these registrations, thus only (i)hospitals having this module and (ii) hospitals willing to participate will be included.

ELIGIBILITY:
Inclusion Criteria:

* Registered maternal request of epidural/spinal anesthesia anesthesia

Exclusion Criteria:

* Not possible to determine gender by first name or by personal knowledge at participating site
* Duplicates
* Misregistered time-points of EDA
* Not receiving EDA (even if the initial intention was to apply EDA)
* Uncertain which anesthesiologist that registered the time-point (more than one anesthesiologist involved in documentation or application)
* None/ambiguous documentation of time-points

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Gender defined by first name
Study Population: All anesthesiologist applying epidurals for labor pain during study time frame
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Time from request of epidural anesthesia to anesthesiologist arrival to labor department | 1minute -24 hours
  The waiting time from midwife request of epidural anesthesia to anesthesiologist arrival

SECONDARY OUTCOMES:
Time from request to application of epidural anesthesia | 1minute-24 hours
  The waiting time from midwife request of epidural anesthesia to anesthesiologist application of epidural anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Johan Lundström, MD,Ph.D, Principal Investigator — Umeå University
Locations (1):
- Centralsjukhuset Kristianstad, Kristianstad, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data can be obtained where no individual could be identified
Supporting Information: Study Protocol, SAP
Time Frame: After study completion
Access Criteria: If appropriate authorities approve of data sharing (Ethical Approval Authority and Swedish Authority for Privacy Protection) data can be accessed

REFERENCES:
- [Background] Jones L, Othman M, Dowswell T, Alfirevic Z, Gates S, Newburn M, Jordan S, Lavender T, Neilson JP. Pain management for women in labour: an overview of systematic reviews. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD009234. doi: 10.1002/14651858.CD009234.pub2. PMID 22419342
- [Background] Barker HM, Simmons SW, Hiscock RJ, Cyna AM, McDonald S. Time to get comfortable with a labour epidural. Anaesth Intensive Care. 2014 Jan;42(1):73-7. doi: 10.1177/0310057X1404200113. PMID 24494256
- [Background] Yurashevich M, Carvalho B, Butwick AJ, Ando K, Flood PD. Determinants of women's dissatisfaction with anaesthesia care in labour and delivery. Anaesthesia. 2019 Sep;74(9):1112-1120. doi: 10.1111/anae.14756. Epub 2019 Jul 1. PMID 31264207
- [Result] Melzack R. The myth of painless childbirth (the John J. Bonica lecture). Pain. 1984 Aug;19(4):321-337. doi: 10.1016/0304-3959(84)90079-4. No abstract available. PMID 6384895